CLINICAL TRIAL: NCT02275455
Title: Design Of WELL Being Monitoring Systems, Application in Autism
Acronym: Do Well B
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-0213; 2014-A00611-46 (Registry Identifier: 2014-A00611-46)
Record Dates: First submitted 2014-10-14; First posted 2014-10-27 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Participants with autism (Experimental)
  Interventions: Behavioral: real life situations
- Aged-matched controls (Experimental)
  Interventions: Behavioral: real life situations

INTERVENTIONS:
Behavioral: real life situations — Four phases will be carried out on autism participants and aged-marched controls: 1) 24-hour baseline pre-experiment (physical activity, sleep), 2) 2-hour in real life situation, 3) 30-minute in a quiet environment, interrupted by a few seconds stressful sound, 4) an interview to get comments and feelings about events that triggered anxiety. Autism and control participants will be together for phases 2 and 3, revealing different physiological responses to the same situations, and thus identifying potentially problematic events.

SUMMARY:
The worldwide prevalence of autism is constantly increasing. People with autisms have difficulties in communication and social interaction resulting from atypical perceptual and information processing, leading to the accumulation of anxiety. Extreme overloading experienced internally may not be visible externally. Identifying stressful situations at an early stage may avoid socially problematic behavior from occurring, such as self-injurious behavior. Activation of the autonomous nervous system (ANS) is involved in the response to anxiety, which can be measured through heart rate variability and skin conductance with the use of a portable device, non-intrusively and pain-free. Thus, developing innovative analysis of signal perception and reaction is necessary, mainly for the non-communicative individuals with autism.

DETAILED DESCRIPTION:
The protocol will take place in real life (home and social environments). We aim to associate modifications of ANS with external events which will all be recorded in a synchrony manner through a specific design (spy glasses with video/audio recording). Four phases will be carried out on autism participants and aged-marched controls: 1) 24-hour baseline pre-experiment (physical activity, sleep), 2) 2-hour in real life situation, 3) 30-minute in a quiet environment, interrupted by a few seconds stressful sound, 4) an interview to get comments and feelings about events that triggered anxiety. Autism and control participants will be together for phases 2 and 3, revealing different physiological responses to the same situations, and thus identifying potentially problematic events. We will apply the statistical analyses developed by our team on continuous ANS data. Detection of abrupt changes will allow segmenting the data in shorter time series of few minutes with a constant mean, and estimating their persistency or antipersistency through a piecewise constant fractal index. We will disentangle classes characterizing different behaviors such as anxiety, rest and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Clear autism spectrum disorder, based on the autism diagnostic interview - revised (ADI-R), the autism diagnostic observation schedule - generic (ADOS-G), and the Vineland adaptive behavior scales (VABS).

Exclusion Criteria:

* change in medical prescription in the previous 3 months and during the experiment.

The same inclusion criteria will apply for the paired age and sex matched individuals with the exception of autism spectrum. The paired control will be chosen within the friends of individuals with autism. In case of difficulty to recruit controls, the psychologist referent may be served as control.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Variability from holter electrocardiogram | at day 1

SECONDARY OUTCOMES:
Heart Rate Variability from the heart rate transmitter belt | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Dutheil, MD PhD, Principal Investigator — University Hospital of Clermont-Ferrand (CHU), France
Locations (1):
- University Hospital of Clermont-Ferrand (CHU), France, Clermont-Ferrand, France, France

REFERENCES:
- [Derived] Dutheil F, Chambres P, Hufnagel C, Auxiette C, Chausse P, Ghozi R, Paugam G, Boudet G, Khalfa N, Naughton G, Chamoux A, Mermillod M, Bertrand PR. 'Do Well B.': Design Of WELL Being monitoring systems. A study protocol for the application in autism. BMJ Open. 2015 Feb 20;5(2):e007716. doi: 10.1136/bmjopen-2015-007716. PMID 25710916
- See also: Related Info — http://math.univ-bpclermont.fr/DoWellB/